CLINICAL TRIAL: NCT03679247
Title: Electronic Tools to Increase Recognition and Improve Primary Care Management for Hypertension in Chronic Kidney Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Lipika Samal, Director of Brigham and Women's Primary Care Practice-based Research Network, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2018P000692; R01DK116898 (NIH)
Record Dates: First submitted 2018-09-11; First posted 2018-09-20 (Actual); Results first posted 2024-11-26 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-11

CONDITIONS: Chronic Kidney Diseases; Hypertension
MeSH Terms: conditions — Renal Insufficiency, Chronic; Hypertension | interventions — Methods

STUDY DESIGN:
Intervention Model Description: Groups of patients sharing the same PCP will be randomized. The groups will be stratified based on two factors (size of group and mean SBP). Within these strata, groups will be randomized to intervention and control arms in a 1:1 ratio. The intervention will be in place for 12 months and data collection will continue for an additional 6 months.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Providers overseeing patients in the intervention arm will receive guidance within electronic health record from clinical decision support system.
  Interventions: Other: Intervention
- Control (Experimental): Providers overseeing patients in the control arm will continue to provide usual care.
  Interventions: Other: Control

INTERVENTIONS:
Other: Intervention — The intervention will be a clinical decision support (CDS) system that contains three main features: 1) methods to synthesize electronic health record (EHR) data in order to identify under-diagnosed chronic conditions (synthesize existing medical data to increase recognition of CKD and uncontrolled HTN in CKD patients and deliver management recommendations based on this evidence), 2) improve the design and content of the CDS using human factors methods, specifically usability testing, and 3) the use of two behavioral "nudges" (pre-checked default orders and an email to obtain commitment from PCPs to obtain their commitment to follow the CDS recommendations).
  Arms: Intervention
Other: Control — Usual Care, PCP will receive an email with general information about CKD guidelines
  Arms: Control

SUMMARY:
In this project the investigators will create computer reminders through user-centered design and will validate the logic using retrospective electronic health record (EHR) data. Then the investigators will test the reminders in primary care clinics to see if they improve treatment of high blood pressure in early chronic kidney disease.

Hypothesis: The mean systolic blood pressure of the chronic kidney disease (CKD) population can be decreased by an intervention with three innovative features: 1) methods to synthesize EHR data in order to identify under-diagnosed chronic conditions, 2) iterative improvement in clinical decision support (CDS) content through human factors methods to maximize the "informativeness" of the CDS, and 3) the use of behavioral economic principles to create behavioral "nudges" internal and external to the CDS.

DETAILED DESCRIPTION:
Specific Aim 1: To develop and validate the intervention. Specific Aim 1a: To develop and validate the CDS that will: 1) synthesize existing laboratory tests, medication orders, and vital sign data; 2) increase recognition of CKD, 3) increase recognition of uncontrolled HTN in CKD patients; and 4) deliver evidence-based CKD and hypertension (HTN) management recommendations.

Specific Aim 1b: To improve the design and content of the CDS, we will use human factors methods, specifically usability testing.

Specific Aim 1c: To develop a "wrap-around" intervention including two behavioral "nudges": 1) pre-checked default orders, and 2) an email to obtain commitment from primary care providers (PCPs) to obtain their commitment to follow the CDS recommendations.

Aim 1a Study Procedures:

Develop Rules for Evidence-based Recommendations for HTN in CKD: The investigators will leverage past work that they have done in a study that delivered recommendations based on national guidelines. An example of one of the rules is to determine whether anti-hypertensive agents have been prescribed but are not at highest potency. If so, the CDS will deliver a recommendation to increase the dosage. The investigators will also include one-click access to recommended orders.

Implementation: Before the start of the trial, the CDS will be moved to the Production environment in "silent mode" where it will record when it would fire, but it will not be displayed to the user. This step will allow us to validate that the rules are accurately identifying patients and producing the correct recommendations through a chart review. The CDS will be activated in the Production environment on the start date of the clinical trial in Aim 2.

Aim 1b Study Procedures:

Usability Test Procedure: Usability testing clinical scenarios will be developed by subject matter experts. Contextual inquiry sessions will be conducted with PCPs and the investigators will ask for feedback on the usability test procedure, as well as content of test scenarios. The goal of Aim 1b is to iteratively improve other important aspects of the CDS that contribute to the overall informativeness of the CDS. The investigators will conduct two rounds of usability testing with PCPs. After each test, the research team and Epic build specialist will make iterative changes to the content of the CDS and layout of information.

Qualitative analysis: Qualitative methods will be employed to analyze the data. The transcripts will be organized by task and participant and then quotes will be identified that illustrate a user expectation, frustration, or misinterpretation of content or functionality.

Aim 1c Study Procedures:

1. Pre-checked, no-action default: The first nudge will be part of the CDS. The investigators will display the CDS with certain options pre-selected.
2. Pledge email to obtain commitment from PCPs to follow the CDS recommendations: As a starting point, we need to ensure that PCPs are aware of the clinical practice guidelines. At the beginning of the study, we will send an advertisement email to all PCPs in the network. In addition, as part of the intervention, we will ask intervention arm PCPs to commit to following the recommendations presented to them in the best practices advisory (BPA), or writing their rationale in the CDS if they choose not to. By clicking a link in an email, the intervention PCP will come to a REDCap survey asking them to type their name to pledge to consider the CDS recommendations provided in our BPAs. The control PCPs will receive a control email without the specific details about the study and without the REDCap link.

Specific Aim 2: To test the effectiveness of the intervention. Specific Aim 2a: To evaluate whether the intervention developed in Aim 1 significantly decreases mean systolic blood pressure in a population of CKD patients with blood pressure > 140/90. They will evaluate the effectiveness of the intervention in a pragmatic, cluster-randomized controlled trial, randomized at the level of the physician. Secondary outcomes will include hypertension-specific process measures, such as treatment intensification.

Specific Aim 2b: To evaluate whether the intervention improves process measures for quality of CKD care including: annual serum creatinine test, and annual urine albumin test.

Specific Aim 2 Study Procedures Please see below for detailed description of the clinical trial.

ELIGIBILITY:
Patients meeting inclusion criteria below will be enrolled.

Inclusion Criteria:

* 18 years or older
* Has visit with PCP at one of the intervention practices during the 2 years before the study period
* Chronic Kidney Disease, defined as two prior estimated glomerular filtration rate (eGFR) 16-59 mL/min/1.73m2 separated by 90 days (as calculated by CKD-EPI) or two prior urine albumin to creatinine ratio (UACR) >30 mg/g separated by 90 days

Exclusion Criteria:

* Patients receiving care from residents in training
* Patients receiving care from physicians only seeing urgent care and walk-in patients
* Patients with a most recent eGFR ≤ 20 or two previous eGFRs within 2 years separated by at least 90 days ≤ 15

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2026 (Actual)
Dates: Start 2021-02-26 (Actual); Primary Completion 2022-10-26 (Actual); Study Completion 2022-10-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lipika Samal, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chen SW, Gannon M, Kilgallon JL, Chay WI, Rubins D, Salmasian H, Dutta S, McEvoy DS, Wu E, Wright A, McCoy A, Samal L. Applying an Empirical Taxonomy to Alert Malfunctions in a Pragmatic Trial for Hypertension Management in Chronic Kidney Disease. Appl Clin Inform. 2025 Oct;16(5):1457-1464. doi: 10.1055/a-2702-6872. Epub 2025 Oct 28. PMID 41151782
- [Derived] Samal L, Chen SW, Lipsitz S, Baer HJ, Kilgallon JL, Gannon M, Dunk R, Chay WI, Fay R, Sainlaire M, Gao C, Wien M, Garabedian PM, Wu E, Salmasian H, Bates DW, Dykes PC, Wright A, McCoy AB. User Actions within a Clinical Decision Support Alert for the Management of Hypertension in Chronic Kidney Disease. Appl Clin Inform. 2025 May;16(3):595-603. doi: 10.1055/a-2554-3969. Epub 2025 Mar 17. PMID 40097147
- [Derived] Samal L, Kilgallon JL, Lipsitz S, Baer HJ, McCoy A, Gannon M, Noonan S, Dunk R, Chen SW, Chay WI, Fay R, Garabedian PM, Wu E, Wien M, Blecker S, Salmasian H, Bonventre JV, McMahon GM, Bates DW, Waikar SS, Linder JA, Wright A, Dykes P. Clinical Decision Support for Hypertension Management in Chronic Kidney Disease: A Randomized Clinical Trial. JAMA Intern Med. 2024 May 1;184(5):484-492. doi: 10.1001/jamainternmed.2023.8315. PMID 38466302
- [Derived] Samal L, Wu E, Aaron S, Kilgallon JL, Gannon M, McCoy A, Blecker S, Dykes PC, Bates DW, Lipsitz S, Wright A. Refining Clinical Phenotypes to Improve Clinical Decision Support and Reduce Alert Fatigue: A Feasibility Study. Appl Clin Inform. 2023 May;14(3):528-537. doi: 10.1055/s-0043-1768994. Epub 2023 Jul 12. PMID 37437601
- [Derived] Kilgallon JL, Gannon M, Burns Z, McMahon G, Dykes P, Linder J, Bates DW, Waikar S, Lipsitz S, Baer HJ, Samal L. Multicomponent intervention to improve blood pressure management in chronic kidney disease: a protocol for a pragmatic clinical trial. BMJ Open. 2021 Dec 22;11(12):e054065. doi: 10.1136/bmjopen-2021-054065. PMID 34937722

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This multiclinic clinical trial, including 15 hospital-based, ambulatory, and community health center-based clinics, occurred from February 2021 to February 2022. All adult patients with a visit to a PCP in the last two years were eligible and those with evidence of CKD and hypertension were included.
Pre-assignment Details: Groups of patients sharing the same PCP panel (PCP or PCP plus a nurse practitioner or physician assistant) were grouped as units. The units were stratified based on two factors (size of unit and mean SBP). Within these strata, units were randomized to intervention and control arms in a 1:1 ratio. While randomization was done at the PCP panel level, data analyses were done at the patient level.
Units Other Than Participants: Group of patients sharing a PCP Panel
Groups:
- Intervention: Patients will receive care from providers who will receive guidance within electronic health record from clinical decision support system.
  Intervention: The intervention will be a clinical decision support (CDS) system that contains three main features: 1) methods to synthesize electronic health record (EHR) data in order to identify under-diagnosed chronic conditions (synthesize existing medical data to increase recognition of CKD and uncontrolled HTN in CKD patients and deliver management recommendations based on this evidence), 2) improve the design and content of the CDS using human factors methods, specifically usability testing, and 3) the use of two behavioral "nudges" (pre-checked default orders and an email to obtain commitment from PCPs to obtain their commitment to follow the CDS recommendations).
- Control: Patients will receive care from providers who will continue to provide usual care.
  Control: Usual Care, PCP will receive an email with general information about CKD guidelines
Period: Overall Study
Arm/Group | Intervention | Control
Started (Data is reported at the patient level (n=2026). Groups of patients sharing the same PCP panel (PCP or PCP plus a nurse practitioner or physician assistant) were grouped as units. The units were stratified based on two factors (size of unit and mean SBP).) | 1029; 87 Group of patients sharing a PCP Panel | 997; 87 Group of patients sharing a PCP Panel
Completed (Data is reported at the patient level (n=2026). Groups of patients sharing the same PCP panel (PCP or PCP plus a nurse practitioner or physician assistant) were grouped as units. The units were stratified based on two factors (size of unit and mean SBP).) | 1029; 87 Group of patients sharing a PCP Panel | 997; 87 Group of patients sharing a PCP Panel
Not Completed | 0; 0 Group of patients sharing a PCP Panel | 0; 0 Group of patients sharing a PCP Panel

BASELINE CHARACTERISTICS:
Groups:
- Intervention: Intervention arm will receive guidance within electronic health record from clinical decision support system.
  Intervention: The intervention will be a clinical decision support (CDS) system that contains three main features: 1) methods to synthesize electronic health record (EHR) data in order to identify under-diagnosed chronic conditions (synthesize existing medical data to increase recognition of CKD and uncontrolled HTN in CKD patients and deliver management recommendations based on this evidence), 2) improve the design and content of the CDS using human factors methods, specifically usability testing, and 3) the use of two behavioral "nudges" (pre-checked default orders and an email to obtain commitment from PCPs to obtain their commitment to follow the CDS recommendations).
- Control: The control arm will continue to provide usual care.
  Control: Usual Care, PCP will receive an email with general information about CKD guidelines
- Total: Total of all reporting groups
Arm/Group | Intervention | Control | Total
Number analyzed (Participants) | 1029 | 997 | 2026
Age, Continuous [Mean (Standard Deviation); unit: years] | 74.2 (0.3) | 75.4 (0.6) | 75.3 (0.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 670 | 553 | 1223
  Male | 359 | 444 | 803
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  race Race: Asian | 24 | 21 | 45
  race Race: Black | 191 | 151 | 342
  race Race: White | 681 | 671 | 1352
  race Race: Other | 79 | 97 | 176
  race Race: Unknown | 54 | 57 | 111
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 1029 | 997 | 2026
systolic blood pressure [Mean (Standard Deviation); unit: mmHg] | 154.3 (14.2) | 153.7 (14.4) | 154.0 (14.3)

OUTCOME MEASURES:

1. Primary Outcome: Change in Systolic Blood Pressure (SBP) From Baseline to 180 Days
Description: Difference in SBP from baseline to 180 days
Time Frame: 180 days
Measure: Mean (95% Confidence Interval); unit: mmHg
Arm/Group | Intervention | Control
Number analyzed (Participants) | 1029 | 997
mmHg | 14.6 [13.1 to 16.0] | 11.7 [10.2 to 13.1]

ADVERSE EVENTS:
Time Frame: 180 days +/- 60 days
Arm/Group | Intervention | Control
All-Cause Mortality (participants affected / at risk) | 15/1029 | 19/997
Serious Adverse Events (participants affected / at risk) | 0/1029 | 0/997
Other Adverse Events (participants affected / at risk) | 0/1029 | 0/997

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-06-22): https://cdn.clinicaltrials.gov/large-docs/47/NCT03679247/Prot_SAP_000.pdf